CLINICAL TRIAL: NCT06938802
Title: Pilot Study of App-delivered Sleep Coaching Among Cancer Survivors and Bedroom Partners
Brief Title: Pilot Study of App-delivered Sleep Coaching Among Cancer Survivors and Their Partners
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005996
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Sleep quality; Psycho-oncology
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep coaching (Experimental): Participants will receive an 8-week sleep coaching program delivered by smartphone/tablet app
  Interventions: Behavioral: Sleep coaching
- Sleep education (Active Comparator): Participants will receive electronic access to educational information about sleep for 8 weeks
  Interventions: Behavioral: Sleep education

INTERVENTIONS:
Behavioral: Sleep coaching — Participants will receive an 8-week sleep coaching program delivered by smartphone/tablet app
  Arms: Sleep coaching
Behavioral: Sleep education — Participants will receive electronic access to educational information about sleep for 8 weeks
  Arms: Sleep education

SUMMARY:
The proposed study will test the feasibility and acceptability of enrolling and retaining cancer survivors and their bedroom partners in a study evaluating digitally delivered behavioral sleep interventions.

DETAILED DESCRIPTION:
Poor sleep is a common issue among cancer survivors that can persist for years and has been linked to increased symptoms (e.g., depression, fatigue), worse quality of life, and worse clinical outcomes like cancer progression and mortality. Partners of cancer survivors also experience poor sleep, but current interventions typically focus on survivors, leaving partners underrepresented. The proposed study will test the feasibility and acceptability of enrolling and retaining cancer survivors and their bedroom partners in a study evaluating digitally delivered behavioral sleep interventions.

ELIGIBILITY:
Cancer Survivor eligibility criteria:

Inclusion Criteria:

1. Diagnosed with any cancer,
2. Completed curative treatment six months to five years before enrolling (excepting ongoing adjuvant endocrine therapy),
3. Score 8 to 14 on the Insomnia Severity Index (ISI)
4. Have a consistent bedroom partner (i.e., sleep in the same bedroom 4 or more nights per week).

Bedroom partner eligibility criteria:

1) No cancer within the past five years

Both survivors and bedroom partners:

Inclusion:

1. Age > or =18 years,
2. Able to speak and read English,
3. Able to provide informed consent,

   Exclusion:
4. No changes in type or dose of prescription sleep medications in the past three months,
5. Not engaged in behavioral sleep treatment for six months prior to enrollment,
6. Not planning to travel across 3 time zones or more during the eight intervention weeks or for the two weeks leading up to study assessments,
7. Not pregnant at enrollment or planning to become pregnant during the study,
8. No diagnosed or suspected psychiatric or medical condition that could interfere with participation,
9. No commitments that would interfere with regular night time sleep patterns (e.g., shift work),
10. No known untreated non-insomnia sleep disorders (e.g., sleep apnea, restless legs syndrome, hypersomnia, circadian rhythm sleep-wake disorder).

Enrolled participants will be allowed to remain in the study even if the other member of their dyad withdraws.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Satisfaction assessed by study-specific survey after the intervention - acceptability | 8 weeks - Immediately after the intervention
  The intervention/study will be deemed acceptable if, on average, participants report satisfaction with the overall program/study as ≥2 on a 0-4 scale.
Feasibility assessed by recruitment and retention rates | Throughout the recruitment period
  The intervention/study will be deemed feasible if 50% of eligible potential participants enroll and 75% of enrolled participants are retained at post-intervention

SECONDARY OUTCOMES:
Change in sleep health from baseline to immediately after the intervention | 8 weeks - Immediately after the intervention
  Participants will complete 8-item short forms of the Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance and sleep-related impairment measures at baseline and immediately after the intervention. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores on PROMIS measures indicate more of the underlying construct.
Change in insomnia symptoms from baseline to immediately after the intervention | 8 weeks - Immediately after the intervention
  Participants will complete 7-item Insomnia Severity Index at baseline and immediately after the intervention. Scores range from 0-28 with higher scores indicating more acute symptoms of insomnia.
Change in symptom burden from baseline to immediately after the intervention | 8 weeks - Immediately after the intervention
  Participants will complete PROMIS scales assessing fatigue, anxiety, and depression at baseline and immediately after the intervention. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores on PROMIS measures indicate more of the underlying construct.

CONTACTS AND LOCATIONS:
Overall Officials: Rina S. Fox, PhD, MPH, Principal Investigator — University of Arizona College of Nursing
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No